CLINICAL TRIAL: NCT04445506
Title: The Effect of the Short-term Use of Systemic Corticosteroids in COVID-19 Patients in Regard to Hospital Length of Stay, Morbidly and/or Mortality.
Brief Title: Short Term Corticosteroids in SARS-CoV2 Patients
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20-027
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-05

CONDITIONS: Corticosteroids; Covid19; SARS-CoV 2; Steroids; Dexamethasone
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV2 patients that received dexamethasone
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 4mg dexamethasone was given to some patients three times daily for 2 days, 2 times daily for 2 days, once daily for 2 days.

SUMMARY:
The investigators reviewed the charts of SARS-CoV-2 patients with pneumonia and moderate to severely elevated CRP and worsening hypoxemia who were treated with early, short-term dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate disease with at least a 30% increase in CRP within 36 hours of admission, and with increasing oxygen requirements.
2. All patients with severe disease with evidence of escalating oxygen requirements
3. The presence of secondary bacterial infections as a probable cause of increasing CRP levels was excluded in all selected patients.
4. Pulmonary embolism and /or cardiac dysfunction were excluded as probable causes of worsening hypoxia in all selected patients.

Exclusion Criteria:

1. All patients on other treatment modalities- Remdesivir and/or Convalescent plasma who showed evidence of clinical improvement as per decrease in CRP levels and/or oxygen requirements were excluded.
2. Patient with associated COPD exacerbation who would benefit from the use of steroids.
3. Patients with Diabetic ketoacidosis, hyperglycemic hyperosmolar state, active concurrent bacterial infections.
4. Patients with history of steroid-induced mania and/or psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years and older with positive SARS-CoV2 test with CRP greater than 50 mg/L and having greater than 2L Oxygen requirement
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Effect on transfers to ICU and escalation of care needing mechanical ventilation | 2 months

SECONDARY OUTCOMES:
Effect on length of stay | 2 months
Change in CRP levels | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Kwame Dapaah-Afriyie, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided